CLINICAL TRIAL: NCT01894347
Title: Prospective Observational Pilot-study for the Evaluation of the Nephro- an Neurotoxicity in the Anti-infectious Therapy With Inhalative Colistin Therapy for Patients With Ventilator-associated Pneumonia (VAP)
Acronym: LOKALE
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Maria Deja, Prof. Dr. med. Maria Deja, Charite University, Berlin, Germany
Other Study IDs: LOKALE
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Infection Resistant to Multiple Drugs
Keywords: Colistin, MDR, inhalative therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tracheal aspirates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colistin inhalative: Adult ICU patients with
  * invasive ventilation with assumed or assured bacteria with an elevated resistance pattern found in a tracheal or bronchial secretion with or without clinical signs of infection
  * indicated colistin co-therapy or eradication-attempt with inhalative colistin (β-Lactam) therapy according to the standard operation procedure (SOP) of the hospital
  Patients included into the study group receive additional TDM, Monitoring of Neuro-and Nephropathology
  Interventions: Other: TDM, Monitoring of Neuro-and Nephropathology

INTERVENTIONS:
Other: TDM, Monitoring of Neuro-and Nephropathology — Therapeutic drug monitoring of serum levels and Monitoring of Neuro- and Nephropathology

SUMMARY:
Multi-Drug resistant pathogens (MDR) are reported worldwide with increasing incidence, especially in intensive care settings.

One of the drugs which are effective against MDRs, is colistin (polymyxin E). This agent has been reintroduced in response to the increase of MDR pathogens and might be used more often in the future. Data on safety regarding the most important side effects are not sufficiently available. l This study evaluates the toxicity in patients who receive aerosolized colistin.

DETAILED DESCRIPTION:
There is growing evidence that patients in the ICU setting have a special risk profile for consecutive colonization and possible infection due to MDR pathogens.

One therapy option is the use of inhalative colistin, as this agent has been demonstrated to be effective against these pathogens. Data on pharmacodynamics or - kinetics are transferred from older studies or from other patient populations. For patients with pulmonary colonization or infection due to an MDR pathogen the systemic resorption of the drug is not known, consequently systemic side effects including kidney or neural damage are not predictable.

This study focus on patients with inhalative colistin therapy and uses therapeutic drug monitoring to determine the rate of systemic resorption of colistin. For the evaluation of neurotoxicity function of peripheral nerves (neve conduction velocity) and of the eighth cranial nerve is monitored. Nephrotoxicity is estimated by creatinine level (-clearance) and the RIFLE criteria.

ELIGIBILITY:
Inclusion criteria:

* invasive ventilated patients (male and female) with assumed or assured bacteria with an elevated resistance pattern found in a tracheal or bronchial secretion with or without clinical signs of infection
* indicated colistin co-therapy or eradication-attempt with inhalative colistin (β-Lactam) therapy according to the standard operation procedure (SOP) of the hospital

Exclusion criteria:

* Consent of the patient or of the patient´s legal representative can´t be obtained soon
* Age < 18 years
* Included within another, prospective clinical antibiotics-study
* Hypersensitivity to colistin or polymyxin B
* Patients with cystic fibrosis
* Present letter of attorney or patient´s provision, which precludes a priori the participation in studies
* Missing consent for storage of pseudonymised data in context of the study
* The patient is in an institution due to a court injunction or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with invasive ventilation and colonization or infection with MDR pathogens
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events (nephro- or neurotoxicity after aerosolised colistin therapy) | 28 days
  Adverse events are measured based on validated criteria:
  1. creatinine-clearance and RIFLE-criteria
  2. Neuromonitoring (nerve conduction velocity, EEG)

SECONDARY OUTCOMES:
Serum concentration of colistin and β-Lactam antibiotics | 3 days
  Colistin-concentration in serum following inhalative therapy (in mg/L) 2 hours and 8 hours of application and in steady state on day 3 of therapy
Serum levels of colistin and β-Lactam antibiotics (e.g. Meropenem)in mg/L | 3 days
  Serum drug levels in mg/L 2hours, 8 hours and 3 days (steady state) after therapy induction

CONTACTS AND LOCATIONS:
Overall Officials: Maria Deja, Prof., Principal Investigator — Charité Universititaetsmedizin Berlin
Locations (1):
- Charité Universitätsmedizin Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Falagas ME, Siempos II, Rafailidis PI, Korbila IP, Ioannidou E, Michalopoulos A. Inhaled colistin as monotherapy for multidrug-resistant gram (-) nosocomial pneumonia: a case series. Respir Med. 2009 May;103(5):707-13. doi: 10.1016/j.rmed.2008.11.018. Epub 2008 Dec 31. PMID 19118994
- [Background] Falagas ME, Rafailidis PI. Nephrotoxicity of colistin: new insight into an old antibiotic. Clin Infect Dis. 2009 Jun 15;48(12):1729-31. doi: 10.1086/599226. No abstract available. PMID 19438398
- [Background] Michalopoulos AS, Karatza DC. Multidrug-resistant Gram-negative infections: the use of colistin. Expert Rev Anti Infect Ther. 2010 Sep;8(9):1009-17. doi: 10.1586/eri.10.88. PMID 20818945
- [Background] Hamer DH. Treatment of nosocomial pneumonia and tracheobronchitis caused by multidrug-resistant Pseudomonas aeruginosa with aerosolized colistin. Am J Respir Crit Care Med. 2000 Jul;162(1):328-30. doi: 10.1164/ajrccm.162.1.9910071. PMID 10903263
- See also: This study initiative is launched by the ABx study group. — http://www.dgai-abx.de